CLINICAL TRIAL: NCT06279611
Title: An Evaluation of LY007 Cell Injection for Recurrent/Refractory CD20 Was Positive Tolerability, Safety, and Efficacy of B-cell Non-Hodgkin Lymphoma in Open, Single-arm Stage I Clinical Research
Brief Title: An Evaluation of LY007 Cell Injection for r/r B-NHL
Acronym: r/r B-NHL
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Longyao Biotechnology Inc., Ltd. (Other)
Collaborators: The First Affiliated Hospital with Nanjing Medical University (Other); Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LY007C1101
Record Dates: First submitted 2024-02-02; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: B-NHL

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LY007 (Experimental): The CAR T cell preparation to be evaluated in this study is LY007, developed and produced by Shanghai Longyao Biotechnology Co., LTD Cell injection. LY007 cell injection is a chimeric antigen receptor targeting CD20 genetically modified using lentiviral vectors (CAR) Autologous T cells are CD20 CAR-T independently developed by Shanghai Longyao Biotechnology Co., LTD., in the CAR facility The independent co-stimulatory signal receptor OX40 was introduced to increase the proliferation and killing function of CAR-T cells. Table of CAR gene The frame comprises the following elements: (1) MSCVEF1α fusion promoter; (2) Single-chain antibody CD20 scFv targeting CD20; (3) CD8 junction and transmembrane region; (4) Intracellular region of 4-1BB; (5) CD3ζ intracellular region; (6) P2A self-shearing peptide; (7) Co-stimulated receptor OX40
  Interventions: Drug: LY007

INTERVENTIONS:
Drug: LY007 — FC and LY007 infusion

SUMMARY:
An evaluation of LY007 cell injection for recurrent/refractory CD20 was positive Tolerability, safety, and efficacy of B-cell non-Hodgkin lymphoma in open, single-arm Phsea I Clinical research

DETAILED DESCRIPTION:
This is a phase I single-arm, open, "3+3" dose escalation study to evaluate the efficacy of LY007 cell injection Safety, tolerability, PK characteristics, PD characteristics, initial efficacy and immunogenicity.

This study plans to enroll approximately 9-18 subjects with relapsed/refractory CD20-positive B-NHL, including DLBCL (inclusive Histological transformation) and TFL. The number of subjects ultimately enrolled depends on the number of DLT observed during the dose escalation phase The number of incremental dose groups prior to DLT and the determination of MTD or clinically recommended dose.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following inclusion criteria to be enrolled in the study:

1. Age 18-70 years old (including 18 years old and 70 years old), regardless of gender;
2. Can understand the study and have signed the informed consent;
3. Expected survival time > 3 months;
4. The American Eastern Oncology Consortium (ECOG) score was 0-1;
5. Cd20-positive B-NHL was confirmed cytologically or histologically according to WHO 2016 criteria These include diffuse large B-cell lymphomas (including histologically transformed forms) and transformed follicular lymphomas (TFL); (For the expression status of CD20, the histological diagnosis of CD20 has been clearly documented in the past Positive subjects (diagnosis within 3 months prior to screening); Subjects without prior records, Pathological specimens provided or collected by our hospital were diagnosed as CD20 positive; Not without a clear record For those who provide or collect specimens, the researchers and sponsors will decide whether to be included according to their medical records);
6. For recurrent or refractory B-cell non-Hodgkin lymphoma, subjects must have at least been treated with anthracene Treatment with cyclodrugs and rituximab (or other CD20-targeting drugs), and have already received them At least two cycles of treatment; Refractory is defined as the best response to the most recent treatment regimen as disease progression, or the last treatment The optimal response of the regimen (at least 2 cycles) was stable disease with a duration of less than 6 months.
7. Does not meet the criteria for autologous hematopoietic stem cell transplantation (auto-HSCT) or is unwilling to perform autologous transplantation Patients with recurrence or progression after blood stem cell transplantation or autologous hematopoietic stem cell transplantation;
8. The venous access required for mononuclear cell collection can be established, and the hemoglobin is ≥70 g/L and neutral Granulocyte ≥ 1.0×109/L, platelet ≥50×109/L, a single nucleus can be performed by the investigator's judgment Cell collection;
9. Evaluable lesions identified according to the 2014 Lugano efficacy evaluation criteria;
10. Organ functions meet the following requirements:

    1. The investigator assessed sufficient bone marrow function to receive lymphocyte clearance chemotherapy;
    2. Serum creatinine ≤1.5× upper limit of normal (ULN) or creatinine clearance (Cockcroft and Gault) > 30 mL/min/1.73 m2;
    3. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3× ULN (ALT and AST in patients with liver metastasis ≤5×ULN);
    4. Total bilirubin ≤2.0 × ULN (for patients with Gilbert's syndrome or lymphoma invading the liver≤3 × ULN);
    5. Lung function: ≤CTCAE grade 1 dyspnea and oxygen saturation of basic finger pulse in indoor air environment Sum degree ≥92%;
    6. Cardiac function: Normal diastolic function, echocardiography or radiation within 1 month prior to enrollment Sexual nuclide active angiography (MUGA) revealed left ventricular ejection fraction (LVEF) ≥ 50%, no clinically significant pericardial effusion. Exclusion criteria Subjects who meet any of the following criteria will not be enrolled in this study

Exclusion Criteria:

Subjects who meet any of the following criteria are excluded from the study:

1. Fully treated cervical carcinoma in situ and a history of other malignant tumors within 5 years prior to screening Adeno-papillary carcinoma, basal cell or squamous cell skin cancer, local front line after radical surgery Except adenocarcinoma and ductal carcinoma in situ after radical surgery;
2. Hepatitis B surface antigen (HBsAg) positive, or Hepatitis B core antibody (HBcAb) positive and peripheral The blood HBV DNA titer was higher than the lower limit. Hepatitis C virus (HCV) antibody positive and HCV RNA titer was higher than the lower limit of detection. Positive for human immunodeficiency virus (HIV) antibodies; Serological test positive for syphilis;
3. Any of the following unstable diseases (including but not limited to) have occurred in the 6 months prior to screening Stable angina pectoris; Cerebral ischemia or cerebral vascular accident; Myocardial infarction; Congestive heart failure (New York Heart Association [NYHA] classification ≥III); Severe cardiac arrhythmia requiring medical treatment Often; After heart angioplasty or coronary stent implantation or heart bypass surgery; mining History of deep vein thrombosis or pulmonary embolism within 6 months prior to cell collection;
4. Lymphoma involving the central nervous system (CNS) only (subjects with secondary CNS lymphoma) Allow to be included);
5. Previous or clinically significant central nervous system history or disease at the time of screening, such as epilepsy, epilepsy Seizures, paralysis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disease, Organic syndrome or mental illness;
6. Active autoimmune disease (including but not limited to systemic lupus erythematosus, dry disease) within 2 years Dryness syndrome, rheumatoid arthritis, psoriasis, multiple sclerosis, inflammatory bowel disease, Hashimoto Thyroiditis, etc., except for hypothyroidism that can only be controlled by hormone replacement therapy);
7. Active or uncontrolled infection requiring systemic treatment within 14 days prior to apheresis;
8. There are active tuberculosis patients in the screening period;
9. During the screening period, there are lymphoma lesions in the lung or gastrointestinal tract that are considered by investigators to be at risk of bleeding Of patients;
10. Was receiving systemic steroid therapy prior to screening and was determined by the investigator to be prolonged during the study period Subjects treated with systemic steroids; Systemic treatment was used within 72 hours before cell transfusion Alcohol-treated subjects (except for inhalation or topical use);
11. Pre-amperectomy CAR-T therapy (except previous CD19-targeted CAR-T therapy) Efficacy was evaluated as disease stable or at any time at 3 months after CD19 CAR-T reinfusion Efficacy evaluation for patients with disease progression) or other genetically modified T cell therapy;
12. Received autologous stem cell transplantation within 6 weeks before anapheresis;
13. Presence of grade ≥2 acute graft-versus-host disease (GVHD) requiring treatment within 4 weeks prior to anaphermology (Glucksberg standard) or generalized chronic GVHD (Seattle Standard) or by researchers Who may need anti-GVHD therapy during the trial;
14. Treatment with alenzumab 6 months before monocyst, or fludarabine or Fludarabine within 3 months before monocyst Cladobine treatment;
15. Received non-lymphocytotoxic cytotoxic chemotherapeutic drugs within 1 week before anapheresis. If it's a single harvest If the former oral chemotherapy drug has passed at least 3 half-lives, it is allowed to be included in the group.
16. Received lymphocytotoxic chemotherapy (e.g. Cyclophosphamide, IFosfamide, benzene) within 2 weeks of preharvest Damustine);
17. Use of other study drugs within 4 weeks prior to anapheresis. But ineffective or disease progression during the trial, and If at least 3 half-lives had passed before the single harvest, they were allowed to be included.
18. LY007 cell injection received donor lymphocyte infusion (DLI) within 6 weeks prior to administration;
19. Received radiotherapy within 6 weeks prior to anapheresis. Disease progression at the subject's radiotherapy site, or other unirradiated areas Only patients with PET positive lesions were eligible for inclusion. If PET is present in other unirradiated sites For positive lesions, radiotherapy for a single lesion was allowed 2 weeks before anapheresis.
20. Acute side effects caused by previous treatment did not recover to grade 1 or below (hematological toxicity and alopecia) Except);
21. The presence of life-threatening hypersensitivity or other intolerance to the drugs used in the study Severe allergies;
22. Any of the following:

    1. Platelet transfusion within 1 week before enrollment;
    2. Red blood cell (RBC) transfusion within 2 weeks prior to enrollment;
    3. Granulocyte macrophage colony-stimulating factor (GM-CSF) was administered during the first 2 weeks of enrollment.
23. Persons who are pregnant or breastfeeding, or who plan to become pregnant within 1 year after cell transfusion, or partners in their cell cycle Male subjects planning pregnancy within 1 year after transfusion;
24. Any situation that the investigator believes will compromise the safety of the subject or interfere with the purpose of the study or cannot be complied with Adhere to the study protocol or other circumstances that are not suitable for inclusion

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-12-25 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose or clinically recommended dose | Day0 to 2year
  No more than 1 out of 6 subjects experienced the highest dose of DLT. At least 6 subjects need to be evaluated at the MTD dose.
Dose limiting toxicity | Day0 to 2year
  Adverse events (AEs) that meet the following criteria and occur within 28 days after the subject receives LY007 cell injection reinfusion will be classified using the ASTCT 2018 standard for CRS and neurotoxicity, while the remaining AEs will be evaluated using the CTCAE 5.0 standard:
  1. Any grade 4 or 5 AE related to LY007 cell injection after treatment, excluding no clinically significant laboratory test indicators;
  2. Any grade 3 AE related to LY007 cell injection that does not improve to ≤ grade 2 within 7 days after treatment, excluding laboratory test indicators with no clinical significance;
  3. Any grade 3 seizures that occur after treatment and cannot be relieved to ≤ grade 2 within 3 days;
  4. Any ≥ level 3 autoimmune toxicity (excluding B cell dysgenesis) that occurs after treatment.
Adverse Events , Serious Adverse Events , Adverse Events of Particular Concern | Day0 to 2year
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0".

SECONDARY OUTCOMES:
PK aspect | Day0 to 2year
  Number of LY007 cells in peripheral blood after LY007 cell administration.
PK aspect | Day0 to 2year
  copy number of CAR gene in peripheral blood after LY007 cell administration.
PD aspect | Day0 to 2year
  The proportion of lymphocyte subtypes in peripheral blood before and after administration of LY007 cell injection;
therapeutic effect | Day0 to 2year
  Objective response rate (ORR) evaluated according to Lugano 2014 criteria (at least 3 after cell transfusion)
Anti LY007 antibody | Day0 to 2year
  The production of anti LY007 antibody (ADA) in serum
The titer of human anti mouse antibody | Day0 to 2year
  the titer of human anti mouse antibody (HAMA) in serum

OTHER OUTCOMES:
Exploratory study endpoint | Day0 to 2year
  The correlation between the above PK parameters and efficacy (CR, PR, SD, PD);CR=complete remission; PR=partial relief; SD=disease stability; PD=disease progression.The correlation between the expression of CD20 in peripheral blood and tumor lymph nodes at baseline and the efficacy (CR, PR, SD, PD).

CONTACTS AND LOCATIONS:
Overall Officials: Zhao Weili, MD, Principal Investigator — Ruijin Hospital, Shanghai Jiaotong University School of Medicine Recruiting Shanghai, Shanghai, China, 200025
Locations (1):
- Ruijin hospital, Shanghai, Shanghai Municipality, China